CLINICAL TRIAL: NCT04557566
Title: A Randomized Controlled Trial of the Eat Breathe Thrive Yoga for Eating Disorder Recovery Online Course
Brief Title: ED Recovery Course Online RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Eat Breathe Thrive (Unknown)
Responsible Party: Principal Investigator, Catherine Cook-Cottone, Principal Investigator, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004821
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Yoga-Based Recovery Course; Control

STUDY DESIGN:
Intervention Model Description: RCT- EBT Yoga-Based Course and Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBT yoga-based eating disorder course (Active Comparator): Yoga for Eating Disorder Recovery online course. This course will be led by certified facilitators via Zoom and offered over the course of four weeks, comprising one two-hour session per week. The course will continue to recruit and enroll participants until sufficient power is reached for the study.
  Interventions: Behavioral: EBT yoga-based eating disorder course
- Control (No Intervention): Wait list control

INTERVENTIONS:
Behavioral: EBT yoga-based eating disorder course — Yoga for Eating Disorder Recovery online course. This course will be led by certified facilitators via Zoom and offered over the course of four weeks, comprising one two-hour session per week. The course will continue to recruit and enroll participants until sufficient power is reached for the study.
  Arms: EBT yoga-based eating disorder course

SUMMARY:
The purpose of this study is to examine whether the Eat Breathe Thrive (EBT) Yoga for Eating Disorder Recovery online course is effective in supporting eating disorder recovery.

DETAILED DESCRIPTION:
We will conduct a block randomized controlled trial (RCT) comparing an intervention group and a waitlist control group. Participants in the intervention group will complete the Eat Breathe Thrive (EBT) Yoga for Eating Disorder Recovery online course. This course will be led by certified facilitators via Zoom and offered over the course of four weeks, comprising one two-hour session per week. The course will continue to recruit and enroll participants until sufficient power is reached for the study. At Pretest, Posttest 1, Posttest 2, and three-months Follow-Up, participants will complete a series of self-report measures (see point 12.3). Participants in the waitlist control group will only be engaged in the study assessment procedures. However, they will be given the opportunity to take part in the Yoga for Eating Disorder Recovery online course that was delivered to the intervention group, once Posttest 1 has been completed by both groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in the study sample will be people between the ages of 18 and 65, who self-identify as women, are not pregnant, are willing to sign the consent form, are English-speakers, have not taken any EBT course before, and self-identify as recovering from an eating disorder.

Exclusion Criteria:

* The study will utilize the EBT participant application for screening (see attached). Further, those excluded will be people who do not self-identify as women, who are below 18 years old or above 65, pregnant, unable/refuse to sign the consent form, non-English speakers, have taken EBT before, and who do not self-identify as recovering from an eating disorder. Further, those who have suicidal ideations and engage in self-harm behaviors cannot be included.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female
Enrollment: 277 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Reduced Eating Disorder Behaviors | at 4, 12, and 24 weeks
  Reduced Eating Disorder Behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, SUNY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No